CLINICAL TRIAL: NCT07287917
Title: A Phase 1b/2 Trial Investigating the Safety and Efficacy of Oral AMXT 1501 and Oral DFMO in Combination With Standard of Care in Patients With Advanced Solid Tumors Who Progressed After Prior Therapies
Brief Title: Study of AMXT 1501 and DFMO in Combination With Standard Therapies in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aminex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMXT1501-103
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Melanoma (Skin Cancer); HER2-low Hormone Receptor Positive Breast Cancer
Keywords: breast cancer; melanoma; AMXT 1501; DFMO; polyamine inhibitor; advanced solid tumor; combination therapy; polyamine
MeSH Terms: conditions — Melanoma; Breast Neoplasms | interventions — Eflornithine; Fulvestrant; capivasertib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Breast Cancer (ER+ HER2-) (Experimental): Arm 1: Breast Cancer Cohort (Cohort 1: ER+ / HER2-)
  AMXT 1501 oral
  DFMO oral
  Fulvestrant IM
  Capivasertib PO
  Interventions: Drug: AMXT 1501 Dicaprate; Drug: DFMO; Drug: Fulvestrant; Drug: Capivasertib
- Arm 2: Melanoma (Experimental): Arm 2: Melanoma Cohort (Cohort 2: Melanoma)
  AMXT 1501 oral
  DFMO oral
  Pembrolizumab IV
  Interventions: Drug: AMXT 1501 Dicaprate; Drug: DFMO; Drug: Pembrolizumab

INTERVENTIONS:
Drug: AMXT 1501 Dicaprate — Formulation: Enteric-coated oral tablet (100 mg base)
  Dose: Body-surface-area-adjusted; starting dose = 300 mg PO BID; may escalate per 3 + 3 design
  Administration: By mouth on an empty stomach (AM and PM doses)
  Other Names: AMXT 1501
Drug: DFMO — Formulation: 500 mg gel capsule
  Dose: 500 mg PO once or twice daily, per cohort dose level
  Other Names: Difluoromethylornithine
Drug: Fulvestrant — Dose: 500 mg IM injection on Day 2 and Day 15 of Cycle 1, then Day 2 of each subsequent 28-day cycle
  Arms: Arm 1: Breast Cancer (ER+ HER2-)
Drug: Capivasertib — Dose: 400 mg PO BID for 4 days on / 3 days off each week (28-day cycle)
  Arms: Arm 1: Breast Cancer (ER+ HER2-)
Drug: Pembrolizumab — 200 mg IV infusion every 3 weeks (Q3W) for up to 12 months
  Other Names: Keytruda®
  Arms: Arm 2: Melanoma

SUMMARY:
This study will evaluate the safety, tolerability, and preliminary effectiveness of AMXT 1501 and DFMO when combined with standard treatments for advanced solid tumors. The trial includes two groups:

* Cohort 1: Patients with ER+ / HER2- breast cancer receiving fulvestrant and capivasertib
* Cohort 2: Patients with unresectable or metastatic cutaneous melanoma receiving pembrolizumab

The Phase 1b portion will find the recommended Phase 2 dose (RP2D). The Phase 2 portion will further evaluate clinical activity at the RP2D using response criteria for solid tumors (RECIST 1.1).

The study will also evaluate pharmacokinetics, pharmacodynamics, disease control, and overall safety.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1b/2 clinical trial evaluating the combination of oral AMXT 1501 and oral DFMO with standard of care (SOC) therapies in patients with advanced solid tumors who have progressed after prior therapy.

AMXT 1501 is a polyamine transport inhibitor, and DFMO is an inhibitor of polyamine biosynthesis. Together, they are designed to reduce tumor polyamines and potentially improve tumor response to standard cancer treatments. Preclinical and early clinical studies suggest that dual polyamine blockade may reduce tumor growth and reverse tumor-induced immunosuppression.

Cohort 1: ER+ / HER2- Breast Cancer

Patients receive AMXT 1501 + DFMO in combination with:

Fulvestrant 500 mg IM

Capivasertib 400 mg PO BID (4 days on, 3 days off)

Cohort 2: Unresectable or Metastatic Cutaneous Melanoma

Patients receive AMXT 1501 + DFMO in combination with:

Pembrolizumab 200 mg IV every 3 weeks

Phase 1b (Safety Run-In)

The primary objective is to evaluate safety, tolerability, dose-limiting toxicities (DLTs), and to identify the recommended Phase 2 dose (RP2D). A standard 3+3 dose-escalation design is used.

Phase 2 (Dose Expansion)

The study evaluates the efficacy of the combination regimens using:

Objective response rate (ORR)

Duration of response (DOR)

Disease control rate (DCR)

Progression-free survival (PFS)

Overall survival (OS)

Pharmacokinetics, pharmacodynamics, and biomarker analyses (including tumor biopsies) will also be conducted.

Up to approximately 92 patients will be enrolled across the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for study participation only if they meet ALL the inclusion criteria applicable to their diagnosis.

1. Understand and sign the informed consent form (ICF) and be willing to comply with all study procedures before any study specific procedures are conducted.
2. ≥18 years old at the time of signing the informed consent.
3. Diagnosed with unresectable, locally advanced, or metastatic solid tumors including ER+ HER2- breast cancer (Cohort 1) or melanoma (Cohort 2)

   a.Underlying malignant disease must be histologically or cytologically documented b.For breast cancer patients: locally advanced or metastatic breast cancer with one or more actionable PIK3CA/AKT1/PTEN-alterations following progression on at least 2 endocrine-based regimens in the metastatic setting or recurrence on or within 12 months of completing adjuvant therapy. Patients who are candidates to start therapy with capivasertib are eligible for enrollment. Patients previously treated with PIK3CA inhibitors will be allowed into the study. Premenopausal patients with ER+ HER2-breast cancer may be enrolled and should be maintained on an agent for ovarian suppression (i.e., luteinizing hormone-releasing hormone [LHRH] agonist) as part of SOC.

   c.For melanoma patients: patients with unresectable metastatic cutaneous melanoma that progressed on any prior immune checkpoint inhibitor and, if BRAF600 mutant positive, a BRAF or mitogen-activated protein kinase (MEK) inhibitor or both as shown below: i.Patient have to have resolution of all immune checkpoint inhibitor-related adverse events to Grade 0-1 and prednisone ≤10 mg/day for at least 2 weeks. Histologically or cytologically confirmed diagnosis of unresectable Stage III or metastatic melanoma not amenable to local therapy.

   ii.Patients must have progressed or shown intolerance to any prior immune checkpoint inhibitors.

   iii.Patients with BRAF gene mutant melanoma must have had a prior treatment regimen (progressed or shown intolerance) that included vemurafenib, dabrafenib, or an approved BRAF gene and or MEK protein inhibitor. However, patients who may continue to be candidates for second line immune check point inhibitors can be enrolled prior to initiation for BRAF gene or MEK inhibitors.

   iv.Patients with incurable malignancies may be enrolled regardless of the number of prior treatment lines, as long as in the opinion of the Investigator, the patient would be unlikely to tolerate or derive clinically meaningful benefit from other available treatment options (FDA Guidance for Industry: Cancer Clinical Trial Eligibility Criteria: Available Therapy in Non-Curative Settings. July 2022).

   d.Has evaluable or measurable disease by tumor Response Evaluable Criteria in Solid Tumors version 1.1 (RECIST 1.1) at the time of enrollment. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   e.Patients with brain previously treated stable brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
4. Patients must be willing to undergo a fresh tumor biopsy at Screening and during treatment if safe and clinically feasible. An archival sample is allowed if obtained within 1 year prior to the first dose of study drug. However, lack of tumor biopsy by itself will not preclude patients from enrollment.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at Screening or Day 1.
6. Life expectancy of at least 12 weeks.
7. Adequate organ function defined as:

   a.Absolute neutrophil count (ANC) ≥1.5×109/L without granulocyte colony-stimulating factor (G-CSF) support within 7 days preceding the laboratory assessment b.Platelet ≥100×109/L, without transfusion within 7 days preceding the laboratory assessment c.Hemoglobin ≥9 g/dL, without transfusion support within 7 days preceding the laboratory assessment d.Activated partial thromboplastin time/partial thromboplastin time (aPTT/PTT) ≤1.5×ULN e.Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (if liver metastases are present, then ≤5×ULN is allowed) f.Total serum bilirubin ≤1.5×ULN, except for patients with known Gilbert's Syndrome in whom ≤3×ULN is permitted. Confirmation of Gilbert's diagnosis requires elevated unconjugated (indirect) bilirubin values; normal complete blood count in previous 12 months, blood smear, and reticulocyte count; normal aminotransferases and alkaline phosphatase in previous 12 months g.The patient is clinically euthyroid (whether treated or untreated) h.Renal: Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min/1.73 m2 for patients with serum creatinine levels >1.5×ULN i.Any Grade 3 or higher laboratory abnormalities should be discussed and approved by the Sponsor Medical Monitor or designee prior to enrollment (even if not considered clinically significant)
8. Fully recovered from acute toxic effects of prior anti-neoplastic therapies. The following minimum periods from treatment apply:

   1. Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
   2. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g., Neulasta) or 7 days for short-acting growth factor.
   3. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.

   The duration of this interval must be discussed with the Sponsor Medical Monitor or designee.

   d.Monoclonal antibodies: >21 days must have elapsed from the infusion of last dose of antibody and toxicity related to antibody therapy must be recovered to Grade ≤1.

   e.Radiation therapy: Patients must have had their last fraction of craniospinal or focal irradiation a minimum of 8-12 weeks prior to enrollment.

   f.Stem cell transplant: Patients must be ≥3 months since autologous stem cell transplant. Patients who received allogenic stem cell transplant or solid organ transplant are not eligible for study.

   g.For combination with pembrolizumab cohort: Patients with Grade ≤2 neuropathy may be eligible, as may patients with endocrine-related Grade ≤2 AEs requiring treatment or hormone replacement.
9. Active secondary malignancies will not be allowed, with the exception of:

   a.Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer b.Adequately treated Stage 1 cancer from which the patient is currently in remission and has been in remission for ≥2 years c.Low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 ng/mL d.Any other cancer from which the patient has been disease-free for ≥3 years
10. Patient compliance and geographic proximity (as determined by the Investigator) to allow adequate follow-up.
11. Both male and female patients must be willing to consent to using highly effective contraception (refer to Section 9.1.10) prior to study entry, while on treatment, and at least 3 months thereafter.
12. Able to take oral medications.

Exclusion Criteria:

Patients will not be eligible for study participation if they meet ANY of the exclusion criteria.

1. Patients with melanoma only:

   i. Radiation therapy, or biological cancer therapy within 4 weeks prior to the first dose of study drug, or not recovered from the AEs due to cancer therapies administered more than 4 weeks earlier ii.Expected to require any other form of systemic or localized antineoplastic therapy while on study.

   iii.Chronic systemic steroid therapy within 2 weeks before the planned date of the first dose of randomized treatment or on any other form of immunosuppressive medication.
2. Intolerant to any component of combination or standard of care therapies.
3. History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. Patient has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
4. Active inflammatory neurological disorders (e.g., Guillain-Barre Syndrome, amyotrophic lateral sclerosis, multiple sclerosis).
5. Treatment with radiation therapy, surgery, chemotherapy, or immunotherapy within 4 weeks prior to study entry (6 weeks for nitrosoureas or Mitomycin C). No prior use of Adriamycin is allowed. Limited prior palliative radiation may be permissible no less than 2 weeks prior to C1D1 with approval from the Sponsor Medical Monitor or designee.
6. Targeted small molecule therapy within 7 days prior to initiation of trial therapy. Chemotherapy within 14 days prior to initiation of trial therapy.
7. Active autoimmune disease (e.g., lupus, rheumatoid arthritis, Sjogren's syndrome) requiring systemic treatment (i.e., disease modifying agents, corticosteroids, or immunosuppressive drugs) in the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. History of or presence of clinically significant cardiovascular disease, e.g.,

   a. Inadequately controlled or uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg on antihypertensive medications.) b. Atherosclerotic cardiovascular disease including history of myocardial infarction, unstable angina, angina, coronary artery disease, cerebrovascular accident (CVA) or transient ischemic attack (TIA). History of coronary revascularization including coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI) or stent placement is excluded. c. Elevated Troponin I or BNP (or NT-proBNP) blood levels above the upper limit of normal at screening or baseline on C1D1.

   d. Heart failure or abnormal left ventricular ejection fraction (e.g., EF <50%).

   e. Atrial or ventricular arrhythmias, including atrial fibrillation, ventricular tachycardia. Patients with pacemakers or ICDs (implantable cardioverter defibrillators) are excluded.

   f. Known cardiac involvement of a systemic disease (e.g., as in SLE, rheumatoid arthritis, psoriatic arthritis, systemic sclerosis
9. History or presence of ECG abnormalities, e.g.,

   a. Congenital or acquired prolonged QTc. Screening QTcF > 450ms is excluded. b. Bundle branch block including right or left bundle branch block, left anterior or posterior fascicular block, second, and 3rd degree AV block, clinically significant ST segment elevations or depressions (e.g., ≥1 mm elevation or ≥0.5 mm depression), arrhythmias. Sinus arrhythmia is not excluded. Asymptomatic sinus bradycardia is not excluded.
10. Had major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1.
11. Have active bacterial, viral, or fungal infections requiring systemic therapy.
12. Women who are pregnant or lactating. NOTE: Women of childbearing potential (WOCBP) must have a "negative" serum pregnancy test within 1 week prior to treatment.

    a.Women not OCBP is defined as: i.Postmenopausal with >1 year since last menses and:

1.If <65 years old, follicle-stimulating hormone (FSH) >40 mIU/mL. 2.If ≥65 years old and not on hormone replacement therapy (HRT), FSH >30 mIU/mL.

3.If ≥65 years old and on HRT, the FSH requirement is not applicable. Postmenopausal females on HRT will be allowed if HRT has been stable for ≥6 months prior to dosing of study drug(s).

4.Written medical documentation of being sterilized (e.g., hysterectomy, double oophorectomy, bilateral salpingectomy) with the procedure performed ≥6 months prior to dosing study drug(s).

Note: Tubal ligation is not considered a form of permanent sterilization. 13.Patients may not have any unresolved toxicity Grade >1 from previous anticancer therapy, except for stable chronic toxicities that are not expected to resolve (i.e., peripheral neuropathy, alopecia, etc.). Patients who have an ongoing requirement for thyroid replacement therapy from prior exposure to an immune checkpoint inhibitor but who are clinically euthyroid are permitted (whether treated or untreated).

14.Have an unwillingness or inability to comply with required procedures in this protocol.

15.Current active liver disease from any cause, including hepatitis A (hepatitis A virus immunoglobulin M [Hep A IgM] positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Patients with HCV with undetectable virus after treatment are eligible. Patients with a prior history of HBV are eligible if quantitative polymerase chain reaction (PCR) for HBV DNA is negative. Note that elevated levels of biotin may interfere with viral serology testing.

16.Have a serious nonmalignant disease that, in the opinion of the Investigator or the Sponsor Medical Monitor or designee, could compromise protocol objectives.

17.Patients who are currently receiving any other investigational agent or who have received an investigational agent within the last 28 days, with the exception of any patient who participated in Study AMXT1501-101A.

18.Known gastrointestinal (GI) disease or procedure that could interfere with the absorption of study drug, including inability to swallow whole capsules or tablets or conditions that may interfere with absorption. The Sponsor Medical Monitor or designee should be contacted for any questions regarding this exclusion criterion.

19.Patients who have exhibited allergic reactions or intolerability to a similar structural compound, biological agent, or formulation as study drugs used in this study, including AMXT 1501, DFMO, and SOC therapies.

20.Use of other hormonal therapies are not permitted during the study in the breast cancer cohort (Cohort 1). Exception: premenopausal women with ER+/HER2- breast cancer should be maintained on an LHRH agonist for ovarian suppression.

21.Use of biotin (i.e., Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 μg. Note: Patients who switch from a high dose to a dose of ≤30 μg/day are eligible for study entry.

22.Uncontrolled, acute, or life-threatening bacteria, viral, or fungal infection. Patients with ongoing use of prophylactic antibiotics, antifungals, or antivirals are eligible if no evidence of active infection, this includes COVID patients.

Exception: Patients with well-controlled HIV (e.g., CD4 >350/mm3 and undetectable viral load) are eligible.

23.Patient has an active or prior history of autoimmune disease. Exception: patients with type 1 diabetes (if stable, well-controlled, and not brittle), vitiligo, hypo- or hyperthyroid disease, or autoimmune alopecia are permitted if the condition does not require immunosuppressive treatment.

24.Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, non-metastatic squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.

25.Combination with pembrolizumab specific additional exclusion criteria:

1. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
2. Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of trial treatment.
3. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
4. Has history of an allogeneic stem cell transplant or a solid organ transplant.
5. Has a history of radiation pneumonitis. (Note: Cannot receive prior radiotherapy within 2 weeks of start of pembrolizumab. Note: Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation [≤2 weeks of radiotherapy] to non-CNS disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | Within 24 months of last patient enrolled
  Number of participants experiencing dose-limiting toxicities as defined in the protocol, including hematologic and non-hematologic toxicities, treatment-related dosing delays, missed doses, or any toxicity leading to discontinuation during the DLT evaluation period.
Incidence, Frequency, and Severity of Adverse Events (AEs) | Within 24 months of last patient enrolled
  Assessment of all treatment-emergent adverse events graded using CTCAE v5.0, including clinical labs, vital signs, ECGs, cardiac biomarkers, and physical examinations, to evaluate the safety and tolerability of AMXT 1501 + DFMO with SOC.
Objective Response Rate (ORR) (Phase 2) | Within 24 months of last patient enrolled
  Proportion of participants achieving a confirmed Complete Response (CR) or Partial Response (PR) per RECIST v1.1 as assessed by the investigator.
Duration of Response (DOR) (Phase 2) | Within 24 months of last patient enrolled
  Duration for which a patient maintains a confirmed objective response per RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Within 24 months of last patient enrolled
  Percentage of participants achieving CR, PR, or Stable Disease (SD) per RECIST v1.1.
Best Overall Response (BOR) | Within 24 months of last patient enrolled
  Best response recorded (CR, PR, SD, or PD) prior to disease progression, based on RECIST v1.1 criteria.
Percentage of Patients With Pseudo-Progression (iRECIST) (Melanoma Cohort) | Within 24 months of last patient enrolled
  Proportion of patients treated with pembrolizumab (melanoma cohort) who demonstrate pseudo-progression based on iRECIST criteria.
Time to Response (TTR) | Within 24 months of last patient enrolled
  Time interval between start of treatment and initial objective tumor response per RECIST v1.1.
Progression-Free Survival (PFS) | Within 24 months of last patient enrolled
  Time from treatment initiation to disease progression per RECIST v1.1 or death from any cause.
Overall Survival (OS) | Within 36 months of last patient enrolled
  Percentage of participants alive at 6 months and 1 year after starting treatment.
Peak Plasma Concentration (Cmax) of AMXT-1501 and DFMO | During Cycle 1 (each cycle is 28 days)
  Maximum observed plasma concentration (Cmax) of AMXT-1501 and DFMO following oral administration.
Trough Plasma Concentration (Cmin) of AMXT-1501 and DFMO | Predose during Cycles 2 and later (each cycle is 28 days)
  Predose (trough) plasma concentrations of AMXT-1501 and DFMO at steady state.
Plasma Concentration-Time Profile of AMXT-1501 and DFMO | Serial sampling during Cycle 1 (each cycle is 28 days)
  Serial plasma concentrations of AMXT-1501 and DFMO collected to characterize the plasma concentration-time profile.

OTHER OUTCOMES:
Change in Immune-Related Gene Expression in Tumor Tissue | From baseline (Screening) to end of Cycle 2 (each cycle is 28 days)
  Change from baseline in immune-related gene expression measured by NanoString analysis in tumor tissue.
Tumor Tissue Concentration of AMXT-1501 and DFMO | At Screening and end of Cycle 2 (each cycle is 28 days)
  Concentration of AMXT-1501 and DFMO measured in tumor biopsy samples.
Tumor Polyamine Levels | At Screening and end of Cycle 2 (each cycle is 28 days)
  Levels of polyamines measured in tumor tissue samples.
eIF5A Hypusination Levels in Tumor Tissue | At Screening and end of Cycle 2 (each cycle is 28 days)
  Levels of hypusinated eIF5A measured in tumor biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Deyaa Adib, MD, Study Director — Aminex Therapeutics, Inc.
Locations (5):
- United States (5):
  - START Cancer Research New York-Long Island, Lake Success, New York
  - Lumi Research, Houston, Texas
  - Laguna Clinical Research Associates, Laredo, Texas
  - START Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists-Fairfax, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
To be determined.